CLINICAL TRIAL: NCT00307515
Title: A Prospective, Randomized, Controlled Evaluation of Fibrin Sealant 2 (FS2) as an Adjunct to Hemostasis for Soft Tissue Bleeding During Retroperitoneal or Intra-Abdominal Surgery
Brief Title: Evaluation of Fibrin Sealant 2 in Retroperitoneal or Intra-Abdominal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Collaborators: OMRIX Biopharmaceuticals (Industry)
Responsible Party: Jonathan Batiller, MBA, Ethicon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400-05-006
Record Dates: First submitted 2006-03-23; First posted 2006-03-28 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Fibrin Tissue Adhesive; Tissue Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Fibrin Sealant 2 (FS2)
  Interventions: Drug: Fibrin Sealant 2 (FS2)
- 2 (Active Comparator): Oxidized Regenerated Cellulose (Surgicel)
  Interventions: Device: Oxidized Regenerated Cellulose (Surgicel)

INTERVENTIONS:
Drug: Fibrin Sealant 2 (FS2) — FS2 Surgical Sealant Kit: Biological Active Component containing Human Fibrinogen 55-85 mg/mL and Thrombin containing Thrombin 800-1200 IU/mL and Calcium Chloride 5.6-6.2 mg/mL
  Other Names: CROSSEAL*; EVICEL*; tissue adhesive
  Arms: 1
Device: Oxidized Regenerated Cellulose (Surgicel) — Commercially available Surgicel used within label.
  Other Names: Surgicel*
  Arms: 2

SUMMARY:
A comparison of fibrin sealant 2 versus Surgicel® as an addition to standard surgical practice in stopping mild to moderate soft tissue bleeding during retroperitoneal or intra-abdominal surgery.

DETAILED DESCRIPTION:
The time it will take to stop bleeding will be measured and compared between patients who are treated with fibrin sealant 2 to those who are treated with Surgicel®.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects requiring non-emergent retroperitoneal or intra-abdominal surgical procedures
* Presence of an appropriate soft-tissue target bleeding site (challenging bleeding site for which topical hemostatic adjuncts might typically be used) as identified intra-operatively by the surgeon
* Subjects must be willing to participate in the study and provide written informed consent

Exclusion Criteria:

* Subjects undergoing emergency surgery
* Parenchymal or anastomotic bleeding sites will not be considered for randomization
* Subjects with any intra-operative findings identified by the surgeon that may preclude conduct of the study procedure
* Subjects with known intolerance to blood products or to one for the components of the study product
* Subjects unwilling to receive blood products
* Subjects with known autoimmune immunodeficiency diseases (including known HIV
* Subjects who are known, current alcohol and/or drug abusers
* Subjects who have participated in another investigational drug or device research study within 30 days of enrollment
* Female subjects who are pregnant or nursing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Hemostatic success within 10 minutes. | Intraoperative

SECONDARY OUTCOMES:
Absence of bleeding at pre-defined time points within 10 minutes | Intraoperative
Incidence of treatment failures | Intraoperative
Incidence of potential bleeding-related complications | 24 hr prior to discharge, Day 7-14
Adverse events | Intraoperative, 24 hr prior to discharge, Day 7-14

CONTACTS AND LOCATIONS:
Overall Officials: James Hart, MD, Study Director — Ethicon, Inc.
Locations (16):
- United States (16):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Miami Research Associates, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - The Iowa Clinic, Des Moines, Iowa
  - St. Agnes Healthcare, Inc., Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cooper University Hospital, Camden, New Jersey
  - Mt. Sinai Hospital, New York, New York
  - GYN Oncology Associates, Syracuse, New York
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital, Houston, Texas